CLINICAL TRIAL: NCT05787275
Title: Effect of Different Types of Diaphragmatic Strengthening Exercises on Diaphragm Muscle Function in Patients With Post Covid Syndrome. A Randomized Control Trail
Brief Title: Effect of Diaphragmatic Strengthening Exercises on Diaphragm Muscle Function in Patients With Post Covid-19 Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Tamer Ibrahim Abo Elyazed, Associate Professor of Physical Therapy, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BeniSuefU3
Record Dates: First submitted 2023-02-25; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Corona Virus Infection
Keywords: Diaphragmatic function; Post Covid; Exercises
MeSH Terms: conditions — Coronavirus Infections; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): received, traditional medical treatment and no exercise
  Interventions: Other: Control
- diaphragmatic positioning group (Experimental): received diaphragmatic strengthening exercises through patient self-positioning in prone on elbows then do diaphragmatic breathing 10-15 min ,twice/day, 7days/ weak
  Interventions: Other: diaphragmatic positioning
- incentive spirometer group (Experimental): received diaphragmatic strengthening exercises through using of incentive spirometer 10-15 min ,twice/day, 7days/ weak
  Interventions: Other: incentive spirometer

INTERVENTIONS:
Other: diaphragmatic positioning — Traditional medical treatment plus diaphragmatic strengthening exercises through patient self-positioning in prone on elbows then do diaphragmatic breathing 10-15 min ,twice/day, 7days/ weak
  Arms: diaphragmatic positioning group
Other: incentive spirometer — Traditional medical treatment plus diaphragmatic strengthening exercises through using of incentive spirometer 10-15 min ,twice/day, 7days/ weak
  Arms: incentive spirometer group
Other: Control — Traditional medical treatment
  Arms: Control

SUMMARY:
The aim of this work is to study the incidence of diaphragmatic dysfunction after COVID 19 infection and the efficacy of different types of diaphragmatic strengthening exercises on diaphragm muscle function.

ELIGIBILITY:
Inclusion Criteria:

* Male and female above 18 years old
* history of probable or confirmed SARS-CoV-2 infection 3 months from the onset of symptoms or at least 2 months from the end of symptoms .

Exclusion Criteria:

* Subjects under 18.
* Patients known to have chronic lung disease .
* Patients known to have neuromuscular disorder.
* Patients known to have diaphragmatic hernia.
* Patients known to have malignancy.
* Patients with clinical evidence of phrenic nerve injury.
* Patients with recent abdominal or thoracic surgery,
* Patients with history of traumatic lesion possibly affecting diaphragm.
* Subjects with severe malnutrition.
* Patients with BMI more than 30

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic thickness | 6 weeks
  Measured by ultrasonography
Pulmonary Function Test | 6 weeks
  MVV

CONTACTS AND LOCATIONS:
Overall Officials: Tamer Abo Elyazed, Principal Investigator — Beni-Suef University
Locations (1):
- Beni-Suef University, Banī Suwayf, Sharq, Egypt

IPD SHARING:
Plan to Share IPD: Yes